CLINICAL TRIAL: NCT07199101
Title: Development of a Multicenter Low-Dose CT Protocol for Children Based on Low-Dose Simulation Technology and Verification by Clinical Randomized Controlled Trial
Brief Title: Multicenter Pediatric Low-Dose CT Protocol: Development and Clinical Verification
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2025-Y-131-D; YGSKL-SHTech-2025-KF01 (Other Grant/Funding Number: State Key Laboratory of Advanced Medical Materials and Devices, ShanghaiTech University)
Record Dates: First submitted 2025-09-18; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Radiation Dose Reduction
Keywords: Tomography, X-ray computed; Child; radiation dose

STUDY DESIGN:
Intervention Model Description: On the RCT trial procedure, Participants will be randomly assigned to the intervention group (adopting the pediatric low-dose CT protocol established based on LDS) or the conventional CT dose group (adopting China's pediatric CT Diagnostic Reference Level protocol) at a 1:1 ratio. A statistician who is not directly involved in the analysis of study results or image evaluation will develop independent randomization schemes for each participating center using the randomized block design, so as to further reduce inter-center bias and ensure the concealment of the allocation scheme.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine dose CT (No Intervention): Participants will undergo a routine dose CT adopting China's pediatric CT Diagnostic Reference Level protocol
- Low dose CT (Experimental): Participants will undergo a low dose CT adopting the pediatric low-dose CT protocol established based on LDS
  Interventions: Radiation: Low dose CT

INTERVENTIONS:
Radiation: Low dose CT — Participants will undergo a low dose CT adopting the pediatric low-dose CT protocol established based on low dose simulation technique.
  Arms: Low dose CT

SUMMARY:
Children are sensitive to ionizing radiation, and there are significant regional variations in current pediatric CT radiation doses. Although there are studies on low-dose CT targeting single lesions, these studies require clear clinical indications and support from advanced equipment, making widespread promotion difficult. The establishment of low-dose CT protocols is mostly experience-based; when radiologists lack confidence in image quality, the credibility of diagnostic reports is compromised. Therefore, the development of low-dose protocols must meet the diagnostic confidence of most radiologists, enable clear visualization of key anatomical structures in clinical practice, and satisfy the requirements for disease diagnosis.

The purpose of this study is to establish a pediatric low-dose CT scanning protocol using Low-dose Simulation of CT (LDS) technology, and conduct a multicenter randomized controlled trial (RCT) in clinical settings to verify the clinical feasibility of this low-dose CT scanning protocol.

ELIGIBILITY:
Inclusion Criteria:

* Aged 0-17 years.
* Pediatric patients for whom a CT examination is deemed necessary by an attending physician.

Exclusion Criteria:

* Parents/guardians refuse to consent to low-dose CT examination.
* Pediatric patients are in critical condition, with no time allocated for explanation of the randomized controlled trial (RCT) protocol.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2650 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the diagnostic performance of CT findings, including the concordance rate with pathological gold standards, other imaging modalities (e.g., MRI), or clinical diagnoses. | From enrollment to the end of treatment at 12 weeks
  With the clinical diagnosis (finally confirmed in pediatric patients after consultation, based on pathology, laboratory tests, other imaging examinations, and clinical characteristics) as the gold standard, determine the concordance rate between CT findings and clinical diagnoses.

SECONDARY OUTCOMES:
To assess discrepancies in subjective image quality ratings among observers, using the Multi-Rater Concordance Correlation (MCRC) statistical method to evaluate the consistency of ratings across different observers. | From enrollment to the end of treatment at 12 weeks
  To analyze differences in diagnostic confidence in images among observers with different years of experience. For CT diagnostic reports showing insufficient diagnostic confidence, the specific criterion is the frequency of descriptive terms indicating low confidence (e.g., "possible," "further examination required," "follow-up review recommended") in the reports.
  To compare differences in radiation doses (CTDI in mSv) between two CT protocols with different dose settings.
  To calculate the radiation dose (CTDI in mSv) difference between the two protocols based on radiation dose data from dose reports.

CONTACTS AND LOCATIONS:
Locations (20):
- China (20):
  - Beijing Children's Hospital, Capital Medical University, National Center for Children's Health, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Medical Center for Capital Children's Health, Capital Medical University, Beijing, Beijing Municipality
  - National Institute for Radiological Protection, China CDC, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Children's Hospital of Chongqing Medical University, National Clinical Research Center for Child Health and Disorders, Ministry of Education Key Laboratory of Child Development and Disorders., Chongqing, Chongqing Municipality
  - Guangdong Women and Children Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Baoding Hospital, Beijing Children's Hospital Affiliated to Capital Medical University, Baoding, Heibei
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan
  - The Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Affiliated Women's Hospital of Jiangnan University, Wuxi, Jiangsu
  - Children's Hospital of Changchun, Changchun, Jilin
  - the First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi
  - Shanghai Children's Medical Center, School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - ShanghaiTech University, Shanghai, Shanghai Municipality
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xu H, Sun QF, Yue BR, Cheng JS, Niu YT. Results and analysis of examination doses for paediatric CT procedures based on a nationwide survey in China. Eur Radiol. 2024 Mar;34(3):1659-1666. doi: 10.1007/s00330-023-10005-7. Epub 2023 Sep 6. PMID 37672054
- [Background] Bosch de Basea M, Thierry-Chef I, Harbron R, Hauptmann M, Byrnes G, Bernier MO, Le Cornet L, Dabin J, Ferro G, Istad TS, Jahnen A, Lee C, Maccia C, Malchair F, Olerud H, Simon SL, Figuerola J, Peiro A, Engels H, Johansen C, Blettner M, Kaijser M, Kjaerheim K, Berrington de Gonzalez A, Journy N, Meulepas JM, Moissonnier M, Nordenskjold A, Pokora R, Ronckers C, Schuz J, Kesminiene A, Cardis E. Risk of hematological malignancies from CT radiation exposure in children, adolescents and young adults. Nat Med. 2023 Dec;29(12):3111-3119. doi: 10.1038/s41591-023-02620-0. Epub 2023 Nov 9. PMID 37946058